CLINICAL TRIAL: NCT02343471
Title: Whey Protein, Postprandial Lipemia and Cardiovascular Disease: Evaluation of the Effect of a Pre-meal of Whey Protein on Postprandial Lipiemia in Subjects With the Metabolic Syndrome and Type 2 Diabetes
Brief Title: The Effect of Whey Protein Consumed as a Pre-meal on Postprandial Lipemia in Healthy and Subjects With Type 2 Diabetes
Acronym: PREMEAL 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ann Bjørnshave, PhD student, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CERN-Premeal3
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-01

CONDITIONS: Healthy; Type 2 Diabetes
Keywords: Whey proteins; Postprandial lipemia; Pre-meal; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Whey Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 20 g whey protein (Experimental): 20 g whey protein dissolved in 200 milliliter (mL) water is consumed as a pre-meal 15 min prior to the main meal. Additionally, 200 mL water is consumed as a part of the main meal.
  Interventions: Dietary Supplement: 20 g whey protein
- Water (Placebo Comparator): 200 milliliter (mL) water consumed as pre-meal 15 min prior to the main meal. 20 g whey protein dissolved in 200 mL water is consumed as a part of the main meal.
  Interventions: Dietary Supplement: 20 g whey protein

INTERVENTIONS:
Dietary Supplement: 20 g whey protein
  Other Names: Brand name: LACPRODAN® SP-9225 Instant (Lot nr.: D150214)

SUMMARY:
Cardiovascular disease (CVD) is one of the most important and frequent causes of death. Postprandial lipidemia (PPL) is an independent risk factor for CVD, besides the traditional risk factors e.g. hypertension, high LDL-cholesterol, family disposition of CVD and type 2 diabetes (T2D). A high PPL is associated with an increased risk of myocardial infarction and stroke. Reduction of increased PPL, as a part of CVD prevention, is therefore pivotal. Especially in groups with increased risk of CVD, like the metabolic syndrome (MeS) and T2D. Identification of a simple diet-related method will possibly result in reduction of CVD in healthy as well as high-risk subjects.

The aim of this project is to investigate the effect whey protein consumed as pre-meal prior to a fat-rich meal on responses of triglycerides and apolipoprotein B48 (ApoB48) in subjects with type 2 diabetes compared to healthy subjects. Secondarily the aim is to study the responses of glucose, insulin, glucagon, amino acids, inflammatory markers, incretins, rate of gastric emptying and metabolomics. Also satiety feeling will be measured.

Investigators hypothesize that whey protein consumed 15 minutes prior to a fat-rich isocaloric meal reduces triglyceride- and ApoB48 responses more in type 2 diabetic subjects compared to healthy subjects.

The investigators research will hopefully contribute to a better understanding of how PPL can be modified in a simple manner. It will promote innovation to the food industry for development and production of healthy food products, which can be applied in the fight against CVD in the background population in general and high-risk people in particular. Thus, the results of this project can impart knowledge of great importance both to the national and international food industry as well as the healthcare systems.

DETAILED DESCRIPTION:
Using a randomised, cross-over design 12 healthy subjects and 12 subjects with type 2 diabetes will consume a test meal prior to a fat-rich meal. The test meals contain 2 different meal types; on where whey protein is consumed as a pre-meal and another where water is the pre-meal. In the second meal type whey protein is instead consumed as a part of the fat-rich meal. Blood samples are collected before consumption of the pre-meal and after consumption of the fat-rich isocaloric meal during 360 minutes. The fat-rich isocaloric meal is a breakfast containing 1043 kcal (15 E% protein, 65 E% fat and 20 E% carbohydrates). The main-meal is composed of white bread, rye bread, butter, cheese (45 %), salami, egg, bacon, milk (1.5 % fat) and coffee (decaffeinated) and should be consumed over 15 min. Visual Analog Scale (VAS) will be used for determination of subjective satiety feeling.

ELIGIBILITY:
Inclusion Criteria - general:

* Weight stable for the last three month.
* BMI<40

Inclusion Criteria for subjects with type 2 diabetes:

* Diagnosed type 2 diabetes (HbA1c > 48 mmol/l)
* Stable dose of Metformin, Sulfonylurea (SU), insulin and SGLT inhibitors are accepted.

Exclusion Criteria - general:

* Type 1 diabetes
* Type 2 diabetes (HbA1c ≥ 48 mmol/L)
* Fasting plasma triglycerides > 5.0 mmol/L
* Blood pressure > 160/100 mmHg
* Cardiovascular, liver, kidney or metabolic disease
* Corticosteroid treatment
* Pregnancy or lactation
* Alcohol or drug abuse
* Legal incapacity

Exclusion Criteria for subjects with type 2 diabetes:

* Treatment with DPP-4 inhibitors, GLP-1 agonists and basal bolus insulin.
* Fasting blood glucose ≥ 14 mmol/l.

Exclusion Criteria for healthy subjects:

* Prediabetes, defined from the WHO criteria (IGF ≥ 6.1 mmol/l).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Effect on triglyceride response of whey protein as pre-meal after a high-fat meal in healthy subjects and subjects with type 2 diabetes measured as incremental Area Under the Curve (iAUC -15 - 360 min). | Prior to the pre meal (-15 min), prior to the main meal (0 min) and 60, 90, 120, 180, 240 and 360 min post main meal
Effect on apolipoprotein B48 of whey protein as pre-meal after a high-fat meal in healthy subjects and subjects with type 2 diabetes measured as incremental Area Under the Curve (iAUC -15 - 360 min). | Prior to the pre meal (-15 min), prior to the main meal (0 min) and 120, 240 and 360 min post main meal

SECONDARY OUTCOMES:
Glucose responses measured as incremental Area Under the Curve (AUC -15 - 360 min) | Prior to the pre meal -15 min, -10 min, prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal
Insulin responses measured as incremental Area Under the Curve (AUC -15 - 360 min) | Prior to the pre meal -15 min, -10 min, prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal
Glucagon responses measured as incremental Area Under the Curve (AUC -15 - 360 min) | Prior to the pre meal -15 min, -10 min, prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal
Glucagon-like peptide 1 (GLP-1) responses measured as incremental Area Under the Curve (AUC -15 - 360 min) | Prior to the pre meal -15 min, -10 min, prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal
Gastric inhibitory peptide (GIP) responses measured as incremental Area Under the Curve (AUC -15 - 360 min). | Prior to the pre meal -15 min, -10 min, prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal

OTHER OUTCOMES:
Responses of the inflammatory marker monocyte chemotactic protein-1 (MCP-1) measured as incremental Area Under the Curve (AUC -15 - 360 min) | Responses of the inflammatory marker monocyte chemotactic protein-1 (MCP-1) measured as incremental Area Under the Curve (AUC -30/-15 - 360 min)
Change in amino acids concentration from baseline to 360 min | Baseline (-15 min), 30, 180 and 360 min
Responses of free fatty acids measured as incremental Area Under the Curve (iAUC -15 - 360 min). | Prior to the pre meal -15 min, -10 min, prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal
Satiety measured as incremental Area Under the Curve (AUC -15 - 360 min) | Prior to the pre meal -15 min, -10 min, prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal
Responses of the inflammatory marker Rantes measured as incremental Area Under the Curve (AUC -15 - 360 min) | Prior to the pre meal -15 min, -10 min, prior to the main meal (0 min) and 15, 30, 60, 90, 120, 240 and 360 min post main meal
Responses of metabolomics measured as incremental Area Under the Curve (AUC -15 - 360 min) in plasma. | Prior to the pre meal (-15 min), prior to the main meal (0 min) and 120, 240 and 360 min post main meal
Responses of metabolomics measured as incremental Area Under the Curve (AUC -15 - 360 min) in urine | Prior to the pre meal (-15 min), and 120 and 360 min post main meal
Responses of satiety visual analog scale (VAS) measured as incremental Area Under the Curve (AUC -15 - 360 min) | Prior to the pre meal (-15 min), prior to the main meal (0 min) and 30, 60, 90, 120, 150, 180, 210, 240, 270, 300 and 360 min post main meal

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Hermansen, Prefessor, Principal Investigator — Aarhus University Hospital